CLINICAL TRIAL: NCT05082948
Title: Migration Rates of Sutured vs Non-sutured Esophageal Stent Placement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: West Virginia University (Other)
Responsible Party: Principal Investigator, Shailendra Singh, Associate Professor & Director, Bariatric Endoscopy, West Virginia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2101223876
Record Dates: First submitted 2021-10-06; First posted 2021-10-19 (Actual); Last update posted 2024-04-23 (Actual); Status verified 2024-04

CONDITIONS: Dysphagia, Esophageal; Esophageal Cancer
Keywords: esophageal stent; dysphagia
MeSH Terms: conditions — Deglutition Disorders; Esophageal Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Suture arm (Experimental): Esophageal stent will be placed in standard of care fashion by the endoscopists using standard gastroscopes. After esophageal stent placement, endoscopic suturing will be performed in cases of patients randomized to suture fixation.
  Interventions: Other: Suture fixation of stent
- Non-suture (Placebo Comparator): Esophageal stent will be placed in standard of care fashion by the endoscopists using standard gastroscopes. No sutures will be placed to fixate the stent
  Interventions: Other: Non suture

INTERVENTIONS:
Other: Suture fixation of stent — Esophageal stent will be placed in the standard of care fashion by the endoscopists using standard gastroscopes. Covered self-expanding metal stent will be placed as per endoscopist preference. After esophageal stent placement, endoscopic suturing will be performed in cases of patients randomized to suture fixation.
  Arms: Suture arm
Other: Non suture — Standard placement of stent without suture fixation
  Arms: Non-suture

SUMMARY:
No standard approach currently exists for endoscopic esophageal stent placement, and both sutured and un-sutured techniques are employed for esophageal stent placement currently. The primary purpose of this study is to find out if suture fixation of esophageal stents is superior to non-suture fixated stent placement.

Consecutive patients who are scheduled for esophageal stent placement will be identified as potential study participants by study personnel and will be approached on the day of the procedure. Informed consent will be obtained and patients will be randomized into suture fixation and non-suture fixation groups. Patients in the suture fixation group will have their esophageal stent secured in location with two endoscopic sutures. Those in the non-suture fixation group will have no sutures placed. Main study outcome is stent migration, and rates of stent migration will be compared in the two groups.

DETAILED DESCRIPTION:
Esophageal stents are commonly placed for both benign and malignant etiologies. Uncovered or partially covered metal stents are employed for malignant conditions while fully covered self-expanding metal stents (FC-SEMSs) are generally placed for the management of benign conditions. FC-SEMSs are also commonly used for managing perforations, fistulae as well as for palliation of symptoms that result from benign structuring disease. Due to the difficulty of uncovered stent removal, FC-SEMSs and partially covered self-expanding metal stents (PC-SEMS) are increasingly utilized for patients with malignancy undergoing neo-adjuvant chemotherapy. Stent migration remains the most frequently encountered complication and the main drawback to their use. While some tissue in-growth is expected in the uncovered metal stents with resulting stability, the silicone coating in covered SEMSs, and to some degree in partially covered stents prevents ingrowth, resulting in higher rates of stent migration; rates exceeding 40% are reported in current scientific literature.2 In recent years, suture fixation of stents has been explored for migration mitigation however data is limited to retrospective series and real-world practice varies depending on endoscopist expertise and experience.

The OverStitch Endoscopic Suturing System (Apollo Endosurgery Incorporation, Austin, TX) is an FDA approved endoscopic suturing system initially designed for closure of gut wall during NOTES procedures,3 however it is now commonly employed for closing perforations, leaks, and has recently garnered attention for stent fixation by suturing in place. At West Virginia University, this device is used, depending on endoscopist preference, to suture esophageal stents to prevent migration. The Investigators aim to perform a randomized clinical trial of endoscopic suture fixated and un-sutured stent placement and compare stent migration rates, technical success, clinical success, and adverse events along with healthcare cost utilization in the two groups.

A randomized controlled trial will be performed at WVU Ruby Memorial Hospital. Patients who are scheduled for esophageal stent placement will be identified as potential study participants by study personnel and will be approached by study personnel on the day of the procedure. Eligibility will be confirmed, and study procedures will be explained. After informed consent is obtained, the patient will be randomized to one of the two groups and the endoscopy will be informed. Each group will consist of 30 patients.

Esophageal stent will be placed in the standard of care fashion by the endoscopists using standard Olympus gastroscopes. 18 to 23 mm covered self-expanding metal stent will be placed as per endoscopist preference. After esophageal stent placement, endoscopic suturing will be performed in cases of patients randomized to suture fixation.

Suture securement of the esophageal stents will be performed using commercially available devices. All endoscopes, and suturing devices will be used in accordance with appropriate Directions for Use (DFU) provided by the manufacturer. The OverStitch Endoscopic Suturing System (Apollo Endosurgery Incorporation, Austin, TX) is an FDA approved endoscopic suturing system that will be utilized in the suture fixation cohort. Standard scope reprocessing will be performed as per institutional protocol after use.

Baseline chest radiographs will be obtained within one week of stent placement. Repeat radiographs to assess the esophageal stents will be obtained at 4-12 weeks after stent placement or in the event of worsening or new symptoms. Chest Xrays will be assessed by attending consultant radiologist and stent positioning will be determined by comparison to local anatomic skeletal landmarks.

All patients will be contacted by the study team by telephone 30 days after procedure to assess for any ongoing symptoms or adverse events. Information on unplanned visits including unplanned emergency department visits or inpatient admissions will also be collected. Electronic health records of patients will be reviewed at 30 days after procedure for obtaining information on unplanned ED visits, or inpatient visits.

ELIGIBILITY:
Inclusion Criteria:

* Able to provide informed consent
* Indication for esophageal stent placement

Exclusion Criteria:

* Presence of any contraindication to esophageal stent placement
* Incarceration
* Inability to tolerate anesthesia
* Pregnant status

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2021-07-20 (Actual); Primary Completion 2023-03-15 (Actual); Study Completion 2023-03-15 (Actual)

PRIMARY OUTCOMES:
Composite of stent migration or total stent dislodgement | 4 weeks
  Stent migration will be defined as stent displacement of 20 mm or more from initial chest Xray. 20 mm has been taken as reference due to some fore-shortening that is expected with the stents, and to account for angulation and measurement related inter-radiograph variability.
  Inability to locate stent on chest radiograph or Esophagogastroduodenoscopy (EGD) will be defined as total stent dislodgement, which will be analyzed separately as well as included in the composite outcome.

SECONDARY OUTCOMES:
Total stent dislodgement | 4 weeks
  Inability to locate stent on chest radiograph or EGD will be defined as total stent dislodgement, which will be analyzed separately as well as included in the composite outcome.
Stent Migration | 4 weeks
  Stent migration will be defined as stent displacement of 20 mm or more from initial chest Xray. 20 mm has been taken as reference due to some fore-shortening that is expected with the stents, and to account for angulation and measurement related inter-radiograph variability.
Technical success | 4 weeks
  Technical success will be defined as successful completion of planned endoscopic deployment of FC-SEMS; defined as correct placement of stent, under endoscopic control, through the stenosis, with the head of the stent more than 1 cm over the stricture
Adverse events | 3 months
  Adverse events that will be noted will include bleeding, infection, perforation, and other unexpected procedure of stent related adverse events
Length of procedure | 4 weeks
  Length of procedure will be defined as the time taken from opening of esophageal stent package to complete withdrawal of scope from the patient's body after completion of procedure

OTHER OUTCOMES:
Cost of procedure | 3 months
  Actual cost of procedure charged
Dysphagia | 3 months
  Dysphagia (as assessed by Watson dysphagia score

CONTACTS AND LOCATIONS:
Overall Officials: Shailendra Singh, Principal Investigator — West Virginia University; Arunkumar Krishnan, Study Director — West Virginia University
Locations (1):
- West Virginia University, Morgantown, West Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Singh S, Maan S, Hadi Y, Agrawal R, Adekolu AA, Cohen EM, Ali FS, Fang W, Markovich B, Krafft M, Thakkar S. Endoscopic suturing to prevent migration of esophageal fully covered self-expandable metal stents: a randomized controlled trial (with video). Gastrointest Endosc. 2025 Oct;102(4):525-535.e4. doi: 10.1016/j.gie.2025.02.037. Epub 2025 Feb 28. PMID 40024292